CLINICAL TRIAL: NCT03222596
Title: The Impact of 4-weeks Mild Exercise Training on Living Quality in Ambulatory and Non-ambulatory Multiple Sclerosis Individuals (EDSS From 0-8) in Motivational and Social Supporting Environment: a Randomized Controlled Trial
Brief Title: The Impact of Exercise Training on Living Quality in Multiple Sclerosis Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Tanja Grubic Kezele, PhD, MD, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 602-01/17-01-147
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Multiple Sclerosis; Fatigue; Mental Status Change; Physical Disability; Physical Activity; Mental Impairment; Quality of Life; Disabilities Psychological; Disability Physical; Pain; Energy Supply; Deficiency; Motivation
Keywords: Quality of Life; Fatigue; Physical Disability; Disabilities Psychological; Pain; Motivation; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected into 2 groups: ambulatory and non-ambulatory (wheelchair) MS individuals that will exercise - group (MSE), with related control group (ambulatory and non-ambulatory (wheelchair) individuals who will not exercise) (MSC). In addition, a group of healthy control subjects without MS (HC) will be evaluated.
  Ambulatory and non-ambulatory group of individuals will exercise under the guidance of a physiotherapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Sclerosis Exercise (Experimental): Ambulatory and non-ambulatory MS individuals that will exercise-group (MSE). Intervention is exercise training.
  Interventions: Behavioral: Exercise training
- Multiple Sclerosis Control (no-Exercise) (No Intervention): Ambulatory and non-ambulatory MS individuals that will not exercise-group (MSC).

INTERVENTIONS:
Behavioral: Exercise training — Exercise programme includes breathing and upper limbs exercises.
  Arms: Multiple Sclerosis Exercise

SUMMARY:
The most common symptom displayed in patients with multiple sclerosis (MS) is a pronounced sense of fatigue that can have negative effect on functional ability and quality of life (QOL).

An important goal of researchers and clinicians involves improving the QOL of individuals with MS, and the exercise therapy represents potentially modifiable behavior that positively impacts on pathogenesis of MS and thus the QOL.

However, the main barrier for its application is low motivational level that MS patients experience due to fatigue with adjacent reduced exercise tolerability and mobility, and muscle weakness. Getting individuals with MS motivated to engage in continuous physical activity may be particularly difficult and challenging, especially those with severe disability or Expanded Disability Status Scale (EDSS 6-8).

Till now, researchers have focused their attention mainly on the moderate or vigorous intensity of exercise and on cardiorespiratory training in MS patients to achieve improvements in daily life quality, less indicating the exercise content, and most importantly, breathing exercises.

In addition, it is investigators intention to make exercise for MS patients more applicable and accessible, motivational and easier, but most important, productive.

Investigators think that MS patients experience more stress with aerobic exercise or moderate to high intensity programme exercise, and can hardly keep continuum including endurance exercise, or treadmill.

Hypothesis:

Investigators hypothesis is that 4-weeks of continuous low demanding or mild exercise programme with specific content and an accent on breathing exercise can attenuate primary fatigue in MS patients, especially in those with more severe disability or EDSS from 6-8, and provide maintenance of exercise motivation. Investigators also propose that important assistant factor for final goal achievement is social and mental support of the exercise group (EDSS from 0-8) led by a physiotherapist. This will help to maintain exercise motivation and finally make better psychophysical functioning, and thus better QOL.

DETAILED DESCRIPTION:
This study will include individuals with multiple sclerosis including all MS types with EDSS from 0-8, who will be practicing at the Multiple Sclerosis Association in Rijeka for a period of 1 month, 2 times a week for 60 minutes per exercise (total 8h).

Participants will be randomly selected into 2 groups: ambulatory and non-ambulatory (wheelchair) MS individuals that will exercise - group (MSE), with related control group (ambulatory and non-ambulatory (wheelchair) individuals who will not exercise) (MSC). In addition, a group of healthy control subjects without MS (HC) will be evaluated.

Ambulatory and non-ambulatory group of individuals will exercise under the guidance of a physiotherapist. Exercise will be carried out sitting on the chairs for all participants, regardless of whether participants are able to walk or not. The practitioner of exercises will first demonstrate and explain each exercise. Participants will be emphasized during exercise to stop exercising if there is tiredness, weakness, pain or any other discomfort.

At the beginning of each exercise session, exercise will be initiated by warming muscles and breathing exercises. Therapeutic and abdominal breathing exercises with extended exhalation will be also conducted. Then follow the exercises of stretching and increasing the movement range of the upper limbs. Participants will work with dumbbells and elastic straps to strengthen the muscles of the upper extremities. In the end of training session, there will be devoted to stretching of the muscle groups involved during exercise.

Each participant involved in the study will undergo the examination through several functional tests at the beginning and up to 4-weeks of the study or exercise, including post-exercise questionnaire for motivation analysis:

1. Assessment of pain level using a "Visual Analogue Scale" for pain (VAS). It is a psychometric response scale or a measurement instrument for subjective characteristics that cannot be directly measured. Here, the participants state their degree of agreement with the facial expression shown with the description of the pain in words, including the appropriate number below the image. VAS for pain is 5 units long, 0 to 5 (0-no pain and 5-hardest possible pain). Since every patient experiences a pain differently, this simple test can evaluate and make it visible.
2. An assessment of the functional independence of daily activities and severity of individuals disability using the "Barthel Index". This test measures the level of independent daily functioning such as feeding, bathing, combing, controlling the bowel, bladder control, transferring from the chair, and mobility and climbing on stairs. This determines the level of disability. The test point to the need for help and care. Score range from 0-100.
3. Evaluation of Quality of Life using the abbreviated version of the "36-Item Short Form Survey" (36-SF). It contains 36 questions including 8 subclasses: physical function, role of constraints due to physical problems, physical pain, general health perception, energy level, social function, the role of limitations due to psychological problems and general mental health. The test time is 10 minutes. The scoring system for the SF-36 is relatively complex and is obtained by summing the results for each sub-base separately. Two summaries can be derived from physical subclasses and psychic subclasses. SF-36 is one of "Multiple Sclerosis Quality of Life Inventory" (MSQLI) and Multiple Sclerosis Quality of Life-54(MSQOL-54) .
4. Grip strength testing with hand dynamometer. It will be measured by hydraulic dynamometer (Jamar, Patterson Medical, USA). The dynamometer handle will be set at position number 2. Measurements will be performed on the dominant and non-dominant hand in the neutral position of the wrist and the elbow joint at 90 º. Each gripe must be maximal (3 in a row) for the mean value.
5. Assessment of cognitive ability using the "Standardized Mini-Mental State Examination" test (SMMSE). SMMSE lasts only 5-10 minutes and is therefore a convenient test to use on multiple occasions.

   SMMSE is effective as a screening test for patients with less cognitive abilities than those without it. In addition, with the help of this test, it is possible to measure changes in the cognitive status that may have been corrected by the intervention.
6. Fatigue estimation using the "Modified Fatigue Impact Scale" (MFIS). It is a modified form of the Fatigue Impact Scale based on data obtained from interviews with MS patients on how tiredness affects their lives. This test gives an assessment of tiredness effects on physical, cognitive and psychosocial functioning and can therefore be treated as 3 separate categories. In full-time MFIS consists of 21 questions. The time to complete is 5-10 minutes and the examinee can solve the test without the help of an interviewer. The total points are obtained by summing all the answers or the additions are made separately by the mentioned categories.
7. Questionnaire upon completion of exercise. The final questionnaire will analyse whether the participants really felt health change after exercise cycle and motivated them in a group under the guidance of a physiotherapist to continue self-exercising at home.

Each participant will be familiar with the research protocol to be implemented in accordance with the Code of Ethics and respecting the principles of the Patient Rights. The investigator will explain the use of the tests. Participants will confirm their participation by signing their consent. Participants voluntarily involved in this research will be provided oral and written consent with the explanation of the possibility of giving up at any time during this study without consequences for their further treatment, guaranteed discretion and anonymity of the obtained data.

Statistical data processing:

The results of the research will be statistically analyzed using a computer program of Version 13 (Sigma Plot Scientific Graphing System, v13.0). Statistical significance will be calculated by non-parametric test for dependent samples and parametric test for dependent samples in cases of normal data distribution. Data will be expressed as mean value ± standard error or as a central value of the median value range. The correlation of the observed changes will be investigated by Spearman's correlation for nonparametric data. Significant statistical changes will be considered at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with multiple sclerosis (EDSS 0-8)
* Ambulatory and non-ambulatory (in wheelchairs)

Exclusion Criteria:

* Individuals with contraindications for exercising
* Individuals with multiple sclerosis with EDSS over 8

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Change of fatigue intensity | baseline, after 4 weeks
  Fatigue estimation using the "Modified Fatigue Impact Scale" (MFIS)
Change of pain intensity | baseline, after 4 weeks
  Assessment of pain level using a "Visual Analogue Scale" (VAS) for pain
Motivation. | baseline, after 4 weeks
  Survey made from questions for subjective self-evaluation of motivation efficiency.
Change of physical abilities and limitations. | baseline, after 4 weeks
  Assessment of the functional independence of daily activities and severity of individuals disability using the "Barthell Index".
Change of mental abilities and limitations. | baseline
  Assessment of cognitive ability using the "Standardized Mini-Mental State Examination" test (SMMSE).
Change of quality of life. | baseline, after 4 weeks.
  Evaluation of Quality of Life using the abbreviated version of the "36-Item Short Form Survey" (36-SF) including physical function, role of constraints due to physical problems, physical pain, general health perception, energy level, social function, the role of limitations due to psychological problems and general mental health.
Change of grip strength. | baseline, after 4 weeks
  Grip strength testing using hand hydraulic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Grubić Kezele, PhD, MD, Principal Investigator — Biomedicine investigations
Locations (1):
- Department of physiology and immunology, Medical Faculty, University of Rijeka, Rijeka, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided